CLINICAL TRIAL: NCT02426047
Title: The Feasibility and Tolerability of Medium Chain Triglycerides as an Adjunct to the Dietary Management of Epilepsy in Women With a Catamenial Seizure Pattern on the Modified Atkins Diet
Brief Title: Medium Chain Triglycerides as an Adjunct to the Modified Atkins Diet for Women With Catamenial Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00038562
Record Dates: First submitted 2015-03-10; First posted 2015-04-24 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Epilepsy; Seizure; Catamenial Epilepsy; Medically Resistant Epilepsy; Medically Resistant Seizures
Keywords: seizures; epilepsy; catamenial; ketogenic diet; modified Atkins diet; intractable epilepsy; medically refractory epilepsy; adult; medium chain triglyceride
MeSH Terms: conditions — Epilepsy; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified Atkins diet plus betaquik® (Experimental): Participants will continue on the modified Atkins diet (with a 20 net grams carbohydrate per day limit) and add betaquik® (a liquid emulsion of medium chain triglycerides) for 10 days per month for 5 months. The days chosen are based on their particular catamenial pattern (there are 3 types that have been identified in the literature).
  Interventions: Dietary Supplement: betaquik®

INTERVENTIONS:
Dietary Supplement: betaquik® — Participants will add betaquik® (a liquid emulsion of medium chain triglycerides) for a 10 day time interval starting 2 days prior to and encompassing the primary catamenial pattern.
  Other Names: betaquik

SUMMARY:
The modified Atkins diet (MAD) has been shown to be effective in treating intractable epilepsy. Approximately 55% of the patients started on the diet are women of childbearing age and women with epilepsy often have a pattern of seizures that correlates with their menstrual cycle, called catamenial epilepsy. The investigators have observed that despite an overall reduction in seizure frequency, some women on the MAD continue to have breakthrough seizures in a catamenial pattern. The investigators hypothesize that women with a history of intractable epilepsy who have been on the modified Atkins diet for at least 3 months and have a catamenial seizure pattern will tolerate and be compliant with the addition of a daily amount of betaquik® (a liquid emulsion of medium chain triglycerides) for a 10 day time interval starting 2 days prior to and encompassing the primary catamenial pattern.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥ 18 years
* Already on the modified Atkins diet for at least 3 months and compliant with treatment
* Catamenial seizure pattern (by Herzog criteria) for at least 2 of the past 3 months (as documented by calendars provided with annotations for seizures and menstrual cycle start and end dates)

Exclusion Criteria (basic exclusion criteria for the modified Atkins diet, so patients should have already been screened for these factors):

* Unwilling to restrict carbohydrates
* Significantly underweight (BMI <18.5)
* Kidney disease
* History of hypercholesterolemia (>300 mg/dl) or hypertriglyceridemia (>200 mg/dl)
* Metabolic or mitochondrial disorder
* Pregnancy
* Lactose intolerance or milk allergy
* Aversion to liquids or inability to eat solid food

Exclusion Criteria (specific to this study):

* Men
* Women who are menopausal or peri-menopausal
* Prior use of betaquik® at any time for any duration
* Already using another ketogenic diet supplement on a sporadic basis (unless the patient is using one daily and is willing to continue doing so for the duration of this study)
* Already using coconut oil specifically for catamenial epilepsy within the month prior to enrollment (okay if patient only using for cooking throughout the month)
* Taking a hormonal contraceptive so that they do not menstruate (e.g. taking active instead of placebo oral contraceptive pills to avoid having a period)
* Anticipated need to adjust anti-epileptic medications within the next 6 months
* Anticipated initiation, change, or discontinuation of a hormonal contraceptive within the next 6 months
* Pregnant or anticipated pregnancy within the next 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Compliance as measured by the percent of time the participants drinks betaquik® averaged over 3 months | 6 months
  The primary outcome measure will be compliance with betaquik® (compared to published compliance of MAD and medium chain triglyceride diets) to demonstrate feasibility. The participant will be considered compliant if they drink the required amount of betaquik® on more than 80% of the prescribed days.

SECONDARY OUTCOMES:
Tolerability (10 point tolerance scale) | 6 months
  Secondary outcome measures will be tolerability of betaquik® based on a 10 point tolerance scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie C Cervenka, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

REFERENCES:
- [Background] Kossoff EH, Rowley H, Sinha SR, Vining EP. A prospective study of the modified Atkins diet for intractable epilepsy in adults. Epilepsia. 2008 Feb;49(2):316-9. doi: 10.1111/j.1528-1167.2007.01256.x. Epub 2007 Oct 5. PMID 17919301
- [Background] Herzog AG, Klein P, Ransil BJ. Three patterns of catamenial epilepsy. Epilepsia. 1997 Oct;38(10):1082-8. doi: 10.1111/j.1528-1157.1997.tb01197.x. PMID 9579954